CLINICAL TRIAL: NCT02418598
Title: A Phase I /II Study of Intra-putaminal Infusion of Adeno-Associated Virus Encoding Human Aromatic L-Amino Acid Decarboxylase in Subjects With Parkinson's Disease
Brief Title: AADC Gene Therapy for Parkinson's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: another clinical study for regulatory approval is planned
Sponsor: Jichi Medical University (Other)
Collaborators: Takara Bio Inc. (Industry); Gene Therapy Research Institution,Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Shinichi Muramatsu, Professor, Jichi Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMU-AAV-AADC-PD
Record Dates: First submitted 2015-04-12; First posted 2015-04-16 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease
Keywords: Adeno-associated virus; Aromatic L-amino acid decarboxylase; AAV-hAADC-2; AAV-2; Gene Therapy; Gene Transfer; Parkinson Disease; Basal Ganglia Disease; Brain Disease
MeSH Terms: conditions — Parkinson Disease; Basal Ganglia Diseases; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort1 (Experimental): The target putamen for AAV-hAADC-2 infusion is identified on MRI image that has been taken prior to the operation, and then subjects will be bilaterally infused with a total volume of 200 µL at a total of 4 sites (2 sites in left putamen, 2 sites in right putamen; 50 µL per site) at a flow rate of 3 µL per minute.
  Interventions: Genetic: Cohort1
- Cohort2 (Experimental): The target putamen for AAV-hAADC-2 infusion is identified on MRI image that has been taken prior to the operation, and then subjects will be bilaterally infused with a total volume of 600 µL at a total of 4 sites (2 sites in left putamen, 2 sites in right putamen; 150 µL per site) at a flow rate of 3 µL per minute.
  Interventions: Genetic: Cohort2

INTERVENTIONS:
Genetic: Cohort1 — AAV-hAADC-2 is administered via bilateral intra-putaminal infusion. The number of vector genomes (vg) administered in this cohort is 3x10^11 vg/subject.
  Arms: Cohort1
Genetic: Cohort2 — AAV-hAADC-2 is administered via bilateral intra-putaminal infusion. The number of vector genomes (vg) administered in this cohort is 9x10^11 vg/subject.
  Arms: Cohort2

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy of intra-putaminal infusion of AAV-hAADC-2 (adeno-associated virus encoding human aromatic L-amino acid decarboxylase) by stereotaxic surgery in patients with advanced Parkinson's disease.

DETAILED DESCRIPTION:
Subjects will be hospitalized and conducted the baseline examination on Day -10. The target putamen for AAV-hAADC-2 infusion is identified on MRI image that has been taken prior to the operation, and then subjects will be bilaterally infused with a total volume of 200 / 600 µL at a total of 4 sites (2 sites in left putamen, 2 sites in right putamen; 50 / 150 µL per site) at a flow rate of 3 µL per minute on Day 0.

After the infusion is complete, the cannula devices will be removed, and the surgical incision will be seamed in accordance with usual trephination. After that, cranial CT scan will be performed so as to confirm whether there are complications such as the occurrence of intracranial bleeding or not. Subjects stay in a hospital for 14 days after infusion of AAV-hAADC-2.

Data and Safety Monitoring Board (DSMB) will be evaluated the safety and efficacy of all subjects at 6 months later assessment in low dose cohort. If there are no events relevant to the discontinuance criteria or moderate to severe adverse events with casual relationship, "Definitely related" or "Possibly related", to AAV-hAADC-2 in this cohort, the study moves to high dose cohort.

At the time of 6 months after the infusion, investigator assesses the treatment effect of AAV-hAADC-2 on the basis of subject diaries, clinical assessment and levodopa requirement dosage. At the same time, investigator assesses a relationship between the dose of AAV-hAADC-2 infused and the amount of intra-putaminal expression by FMT-PET imaging.

The investigator also assesses the safety for 5 years after the baseline examination. Long-term follow up study is additionally conducted for 10 years in reference to guideline of FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with idiopathic Parkinson's disease meet diagnostic criteria for Specified Disease designated by the Ministry of Health, Labour and Welfare (1995) : the Research Committee of CNS Degenerative Disease, L-Dopa is effective in the early disease stage and no findings suggestive of CNS Degenerative Disease are found.
2. Age ≤ 75 years at the time of medical treatment.
3. Age at onset ≥ 35 years.
4. Duration of L-dopa therapy ≥ 5 years.
5. Hoehn and Yahr Stage IV in OFF state at the onset of medical treatment.
6. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Scale Part III (MDS-UPDRS-III), minimum motor score of 30 to a maximum motor score of 100 in OFF state.
7. Positive response to dopaminergic therapy as evidenced by remarkable improvement in MDS-UPDRS-III motor score between the defined "OFF" and "ON" state: a minimum 16 points improvement in the MDS-UPDRS-III after dopaminergic therapy.
8. Patients who can undergo the stereotaxic surgery for Parkinson's disease due to the intolerable motor complication minimum score of 4 to a maximum score of 9 in the MDS-UPDRS-IV part B (diurnal fluctuation of symptom) , not responsive to optimal medical therapy.
9. To be able to comply with the requirements, including the frequent clinical examination after medical treatment, in this study.
10. To keep the therapeutic medicine for Parkinson's disease for at least 2 months prior to participation in this study.
11. Written informed consent.

Exclusion Criteria:

1. Patients who is suspected secondary / atypical parkinsonism based on the medical history of cerebral vascular disease, exposure to antipsychotic or toxic agents, and encephalitis or based on the symptom of Progressive supranuclear palsy, Pyramidal tract sign, autonomic sign, Dementia, Hallucination, Delusion and so on or based on the finding by magnetic resonance imaging (MRI) such as Lacunar infarct or atrophy of the midbrain tectum and atrophy of the pons and the cerebellum.
2. Patients with history of 3 hours or more of intensive or violent dyskinesias in the past 6 months.
3. Patients with previous the stereotaxy for Parkinson's disease (pallidotomy, thalamotomy, deep brain stimulation) .
4. Mini-Mental State Examination (MMSE) ≤ 20 or patient with a diagnosis of dementia in the neuropsychological evaluation.
5. Patients with medical history of Hallucination, Delusion, schizophrenia or affective disorder within 6 months of informed consent.
6. Patients with history of significant cardiovascular disease including cerebrovascular accident.
7. Malignant neoplasm in the brain, clinically significant neurological disease (for example significant brain atrophy not consistent with age).
8. History of other malignancy, with the exception of treated carcinoma cutaneum, within 5 years.
9. Uncontrolled hypertension: systolic blood pressure ≥ 160 mmHg.
10. Coagulopathy or need for anticoagulant therapy.
11. Clinically significant immune dysfunction (for example, the case who require the use of immunosuppressive drugs).
12. Geriatric Depression Scale (GDS) short scale ≥ 10 points, or if on antidepressant, the score > 5 points.
13. On monoamine oxidase (MAO)-A inhibitors, or antipsychotic medications.
14. Unable to scan MRI.
15. Cases without abnormal finding in FMT-PET.
16. Premenopausal female or male who desire impregnating a female (excluded: in case when sperm is cryopreserved prior to gene therapy and child is born by using the sperm).
17. Past medical history of convulsive seizure within 3 years or receiving antiepileptic drug or patients with epileptic aberrance in the electroencephalography.
18. Past medical history of serious drug allergy.
19. Patients who have participated in other clinical trial within 6 months.
20. Patients who meet any of the following criteria:

    1. Serious renal disorder ( Cr ≥ 2.0 mg/dl and BUN ≥ 25mg/dl)
    2. Serious hepatic disorder ( AST (GOT) / ALT (GPT) ≤2.5xupper limit of normal (ULN)
    3. Serious diabetes (casual blood glucose or fasting blood glucose ≥ 200 mg/dl and HbA1c ≥ 9 %)
21. Any other patients judged by investigators to be inappropriate for the subject of this study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
The safety of intra-putaminal infusion of AAV-hAADC-2 as measured by adverse events (including Abnormal laboratory test results) with Classification criteria for severity of adverse reactions (dated 29th Jun,1992). | 6 months
  Confirm the adverse events (including Abnormal laboratory test results) with Classification criteria for severity of adverse reactions (dated 29th Jun,1992).

SECONDARY OUTCOMES:
The treatment effect of intra-putaminal infusion of AAV-hAADC-2 | 6 months
  Assess the improvement of Parkinson's symptom as recorded in the subject diaries, clinical assessment and requirement dosage of levodopa.
The amount of intra-putaminal expression of AAV-hAADC-2 | 6 months
  Assesses a relationship between the dose of AAV-hAADC-2 infused and the amount of intra-putaminal expression by FMT-PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Shin-ichi Muramatsu, MD, PhD, Study Chair — Division of Oriental Medicine, Center for Community Medicine, Jichi Medical University; Division of Genetic Therapeutics, Center for Molecular Medicine, Jichi Medical University; Division of Neurology, Department of Medicine, Jichi Medical University
Locations (1):
- Jichi Medical University, Shimotsuke, Tochigi, Japan